CLINICAL TRIAL: NCT05553015
Title: A Real-World Registry Investigating TReprostInil sodiUM in Pulmonary Hypertension (Re-TRIUMPH)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: TReprostInil
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Hypertension; Medication Therapy Management
Keywords: Pulmonary hypertension; Trepostinil sodium
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PH Patients receiving treprostinil sodium treatment: Patients with pulmonary hypertension receiving treprostinil sodium treatment

SUMMARY:
A Real-World Registry investigate Treprostinil sodium used in patients with Pulmonary Hypertension (Re-TRIUMPH).

DETAILED DESCRIPTION:
This study is a multicenter, prospective, single-arm, observational, real-world study conducted in China. Patients who are at least 18 years of age, have been diagnosed with pulmonary hypertension (PH), agree to participate and meet the eligibility requirement will be enrolled in 20 pulmonary vascular centers across the country for the medically reasonable use of intravenous (or subcutaneous) Treprostinil injections. In the event that eligible patients are enrolled in the study, all aspects will be carried out in an observational manner, and no additional methods or procedures will be necessary. The patient and the physician will jointly determine the clinical management of the patient, including the length of treatment. Patients will be followed up for an observation period of at least 1 year. As part of standard clinical practice, patient data will be collected at the first appointment and every three to six months thereafter. After one year of follow-up, data collection will cease.The main purpose is to evaluate the efficacy and adverse reactions of subcutaneous (intravenous) prostacyclin in the treatment of pulmonary hypertension under current clinical practice. The secondary objectives is to understand the drug treatment plan of treprostinil in clinical practice of patients with pulmonary arterial hypertension in China and to understand the efficacy and adverse reactions of treprostinil in the treatment of patients with different types of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary hypertension who consent to receiving Treprostinil injection;
* Patients who must be over the age of 18;
* The informed consent form must be signed.

Exclusion Criteria:

* Patients who have received Treprostinil Injection for less than two weeks;
* Patients who have used Treprostinil within the past three months;
* Any situation that the investigator believes could affect the interpretation of the study results or pose a risk to patients using Treprostinil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension receiving treprostInil sodium treatment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year transplant event-free survival in patients with pulmonary hypertension | 1 year
  1-year transplant event-free survival in patients with pulmonary hypertension

SECONDARY OUTCOMES:
Incidence of adverse events | 1 year
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD#PhD, Study Director — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (1):
- Center of pulmonary vascular disease, Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No